CLINICAL TRIAL: NCT00862212
Title: Phased Treatment for Social Anxiety Disorder and Coping Behaviors in a Medical Setting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Sarah Book, Prinicpal Investigator, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R01AA013379-05A1 (NIH)
Record Dates: First submitted 2009-03-13; First posted 2009-03-16 (Estimated); Last update posted 2013-04-23 (Estimated); Status verified 2013-04

CONDITIONS: Social Anxiety Disorder; Alcohol Use Disorders
Keywords: anxiety; social anxiety; social anxiety disorder; coping behaviors; alcohol abuse
MeSH Terms: conditions — Phobia, Social; Alcoholism; Anxiety Disorders | interventions — Ethanol; Methods

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Brief Alcohol Intervention (Experimental): Half of the subjects will be randomly assigned to receive a brief physician-delivered alcohol intervention designed by the NIAAA to be delivered by primary care and mental health providers.
  Interventions: Behavioral: Brief Alcohol Intervention
- Control Group (No Intervention)

INTERVENTIONS:
Behavioral: Brief Alcohol Intervention — At the Week 6 visit, all subjects who are randomized to the Experimental Group will receive the experimental brief alcohol intervention. The intervention will be in addition to a standard 20-minute physician visit, for a maximum of 30 minutes. The physician will use the Updated NIAAA Clinician's Guide to ask about drinking and will draw the connection between social anxiety and drinking and how they relate to each other. Subjects will be asked to consider making changes in their drinking and if they agree, a goal will be set and progress toward that goal will be monitored at subsequent visits.
  Other Names: Helping Patients That Drink Too Much, NIAAA Guide
  Arms: Brief Alcohol Intervention

SUMMARY:
The purpose of this study is to treat individuals with social anxiety disorder with a Food and Drug Administration-approved medication for the treatment of social anxiety disorder, the antidepressant paroxetine, and to evaluate the impact of an intervention designed to help those individuals cope with anxiety without the use of common coping behaviors.

DETAILED DESCRIPTION:
Psychiatric and alcohol use problems co-occur in a significant number of individuals seeking treatment in mental health treatment settings. However, there is a paucity of research to guide clinical practice. This is especially true for psychiatrists treating patients with anxiety disorders who also present with co-occurring hazardous drinking. If alcohol is being used as a coping strategy, as it is frequently in individuals with social anxiety, it follows that successful treatment of the social anxiety should resolve dysfunctional drinking. However, results from our study completed during the current funding period did not support this hypothesis and suggested, instead, that additional intervention for hazardous drinking is necessary. The proposed project is a natural "next step" in this line of research, and the design and methods are guided and informed by the results our previous work as well as by recently-collected preliminary data. The proposed study will evaluate the phased approach to the treatment of these co-occurring disorders. Social anxiety will be treated first, then, in the Experimental group, the physician will introduce a brief alcohol intervention at a standard time in the course of social anxiety treatment. The hypothesis being tested is that drinking will decrease more in the Experimental group than in the Control group, where only the social anxiety is treated and discussed. The design of the study follows from the results of the project completed in the previous funding period. The intent of the design was to balance scientific rigor with real-world practicality. Individuals who are specifically seeking treatment for social anxiety and who also drink at hazardous drinking levels will be recruited from the community from two treatment sites, one in South Carolina and one in Minnesota. All subjects in the trial will receive 22 weeks of flexible dosing with paroxetine, an FDA-approved medication for the treatment of social anxiety shown to be effective in our previous trial. Half of the subjects will be randomized to receive at Week 6, in addition to routine social anxiety treatment, a brief physician-delivered alcohol intervention following the Updated NIAAA Clinical Guide for Helping Patients Who Drink Too Much. Research assessments will coincide with physician visits and will also include 34 and 46-week post-treatment follow-up visits. The study is a novel test of the phased treatment model, is one of the first studies to address the treatment of co-occurring anxiety and hazardous drinking in a mental health treatment setting, and uses both social anxiety and alcohol interventions that are easily adoptable in real-world mental health clinical practice. If the hypothesis is supported, the study has broad implications for treatment of other co-occurring anxiety and mood disorders and hazardous drinking.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65.
* Meets DSM-IV criteria for Social Anxiety Disorder, generalized type.
* LSAS score greater than or equal to 60.
* Reports drinking at least 15 standard drinks/week or 5 standard drinks/drinking day for men, and at least 8 standard drinks/week or 4 standard drinks/drinking day for women in the past 30 days.
* AUDIT score between 8 and 15 inclusive for men and 4 and 15 inclusive for women.
* Reports no prior medical alcohol detoxification or formal alcohol treatment including regular attendance at self-help groups.
* Treatment seeking for relief of social anxiety, not for alcohol problems.
* Endorses drinking to cope with anxiety at least 40% of the time during or before a social situation, using the Drinking to Cope survey.
* Able to provide informed consent and fill out self-rating forms in English.

Exclusion Criteria:

* Drug dependence in the past 90 days on any drug besides caffeine or nicotine.
* Lifetime diagnosis of bipolar disorder or schizophrenia.
* Significant suicide risk as assessed by the SCID.
* Current use of psychotropic medications.
* Pregnancy, nursing or refusal to use effective birth control if female.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2009-01; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
alcohol use, as indexed by (1) Drinks per Week and (2) Drinks per Drinking Day | 22 weeks

SECONDARY OUTCOMES:
alcohol intervention effect on hazardous drinker status | Weeks 6-22

CONTACTS AND LOCATIONS:
Overall Officials: Carrie L Randall, Ph.D., Principal Investigator — Medical University of South Carolina; Matthew Kushner, Ph.D., Principal Investigator — University of Minnesota
Locations (2):
- United States (2):
  - University of Minnesota, Minneapolis, Minnesota
  - Medical University of South Carolina, Charleston, South Carolina